CLINICAL TRIAL: NCT04096118
Title: Relationship Between Lymph Node Ratio and Survival Rate in Preoperative Chemoradiation Rectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/426
Record Dates: First submitted 2019-04-17; First posted 2019-09-19 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Lymph node after neoadjuvant rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Colorectal cancer is the most-common cancer of the gastrointestinal tract. The number of positive lymph nodes and total number of lymph nodes retrieved are important prognostic factors. In patients who do not receive preoperative chemoradiation, the total number of lymph nodes should be more than 12 nodes to predict accurate staging. In cases of locally-advanced rectal cancer when patients receive neoadjuvant chemoradiation it is sometimes impossible to retrieve adequate amount of lymph nodes due to the chemoradiation effect. Therefore, this study was to evaluate and predict survival rates based on positive lymph node ratio.

DETAILED DESCRIPTION:
The primary endpoint of this study was to assess the lymph node ratio as another predictor for survival rate in preoperative chemoradiation rectal cancer patients. The other secondary objective was to determine the relationship between total harvested lymph nodes and survival rate in each stage. This is a retrospective, single-centered study, collecting data of patients from January 2011 to December 2017. Including a total of 163 patients with rectal cancer who underwent surgery following neoadjuvant chemoradiation. Using Cox regression and Kaplan-Meier survival analysis to determine whether the lymph node ratio can be used to predict the survival rate and determine the cut-off value to distinguish the prognosis of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rectal cancer who underwent surgery following neoadjuvant chemoradiation.
* Patients have tissues confirmed by Pathology
* no metastasis before surgery

Exclusion Criteria:

* Distant metastasis during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with rectal cancer who underwent curative surgery following neoadjuvant chemoradiation.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Survival rates | 5 year
  survival rate in preoperative chemoradiation rectal cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Chairat Supsamutchai, MD, Study Chair — Ramathibodi Hospital; Tanet Chatmongkonwat, MD, Principal Investigator — of Medicine Ramathibodi Hospital, Mahidol University.
Locations (1):
- Chairat Supsamutchai, Bangkok, Bankok, Thailand

IPD SHARING:
Plan to Share IPD: No